CLINICAL TRIAL: NCT04974190
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy of Lavandula Angustifolia Containing Nasal Spray Medical Device in Preventing Deterioration of COVID-19 in Symptomatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Grasses of Eden Ltd (Industry)
Collaborators: Sherutei Briut Clalit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0037-21-COM1
Record Dates: First submitted 2021-07-21; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A control group is allocated a placebo solution
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with actual device with actual solution (Active Comparator)
  Interventions: Device: Nasal Spray Device
- Patients treated with actual device with placebo solution (Placebo Comparator)
  Interventions: Device: Nasal Spray Device

INTERVENTIONS:
Device: Nasal Spray Device — A Nasal Spray apparatus containing a liquid

SUMMARY:
A Nasal Spray device containing Dead Sea minerals and plant extracts, used to shorten duration and mitigate effects of Covid-19 infection in mild to moderate adult patients

DETAILED DESCRIPTION:
A Nasal Spray device containing Dead Sea minerals and plant extracts, designed to incur a PPAR-alpha agonistic effect, used to shorten duration and mitigate effects of Covid-19 infection in mild to moderate adult patients

ELIGIBILITY:
Inclusion Criteria: Having tested positive to Covid-19 on PCR test -

Exclusion Criteria: Pregnancy Low blood pressure On immune system suppressing medications

-

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Covid-19 infection self-testing on days 2, 4 following testing positive on PCR test | First 7 days after testing positive on PCR test
  Testing using a self testing kit of the Quidel QuickView type
Symptoms monitoring | First 7 days after testing positive on PCR test
  Monitoring any disease symptoms reported by patient

IPD SHARING:
Plan to Share IPD: No